CLINICAL TRIAL: NCT00102778
Title: A Phase IIb, 96 Week, Randomized, Open-label Multicenter, Parallel Group, Repeat Dose Study to Evaluate the Safety, Tolerability, PK and Antiviral Effect of Different Doses and Regimens of GW873140 in Combination With Kaletra (Lopinavir and Ritonavir) in HIV-1 Infected Antiretroviral Therapy naïve Subjects
Brief Title: GW873140 In Combination With Kaletra In HIV Infected Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100136
Record Dates: First submitted 2005-02-01; First posted 2005-02-02 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Infection, Human Immunodeficiency Virus I; HIV Infection
Keywords: HIV infected; therapy-naive subjects
MeSH Terms: conditions — Infections; HIV Infections | interventions — aplaviroc; lopinavir-ritonavir drug combination; Lopinavir; Ritonavir

INTERVENTIONS:
Drug: GW873140
Drug: Kaletra (lopinavir/ritonavir)
  Other Names: GW873140

SUMMARY:
This study is a 96-week study designed to evaluate the safety and efficacy of GW873140 in combination with Kaletra in HIV infected, untreated subjects.

DETAILED DESCRIPTION:
A Phase IIb, 96 week, randomized, open-label, multicenter, parallel group, repeat dose study to evaluate the safety, tolerability, pharmacokinetics and antiviral effect of different doses and regimens of GW873140 in combination with Kaletra (lopinavir and ritonavir) in HIV-1 infected antiretroviral therapy naive subjects

ELIGIBILITY:
Inclusion criteria:

* HIV infected, therapy-naive subjects.
* Females must be of either non-childbearing age, or have a negative pregnancy test.
* All subjects participating in this study should be counseled on the practice of safe sex using a proven double barrier method of contraception throughout the study.
* Screening lab result of plasma HIV-1 RNA greater than or equal to 50,000 copies/mL and CD4 cell count greater than or equal to 100 cells/mm3.
* Have CC Chemokine Receptor5-tropic (R5-tropic) or CC Chemokine Receptor5/CXC Chemokine Receptor4-tropic (R5/X4-tropic) virus based on viral tropism test at screening visit.
* Be treatment-naive, defined as less than or equal to 2 weeks of treatment with a protease inhibitor (PI) or an nucleoside reverse transcriptase inhibitor/nucleotide reverse transcriptase inhibitor (NRTI/ NtRTI), or less than or equal to 7 days of therapy with a non-nucleoside reverse transcriptase inhibitor (NNRTI).
* Prior treatment with any entry inhibitor, attachment inhibitor, or fusion inhibitor (experimental or approved) is not allowed.
* Be able to understand and follow with protocol requirements, instructions and protocol-stated restrictions.
* Signed and dated written informed consent prior to study entry.

Exclusion criteria:

* No detection of CXC Receptor4-tropic (X4-tropic) virus only, based on viral tropism test at screening.
* No active Class C AIDS-defining illness.
* No laboratory abnormalities at screen.
* No significant blood loss prior to study start.
* No pregnant or breastfeeding women.
* Additional qualifying criteria to be determined by the physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175
Dates: Start 2004-12; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To select a GW873140 dose and dosage regimen for further evaluation based on comparison of the short-term antiviral activity, safety and tolerability of different oral doses of GW873140 in combination with LPV/r in HIV-1 infected therapy-naive subjects.

SECONDARY OUTCOMES:
HIV-1 RNA decay rate Long-term safety Effects on plasma viral tropismViral resistance to GW873140 and other on-study drugsPK parameters of GW873140 in subjects receiving combination therapy.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (56):
- United States (26):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Bradenton, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Santa Fe, New Mexico
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Hampton, Virginia
- Canada (5):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Sainte-Foy, Quebec
- Denmark (2):
  - GSK Investigational Site, Copenhagen
  - GSK Investigational Site, Hvidovre
- France (7):
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Denis
  - GSK Investigational Site, Tourcoing
  - GSK Investigational Site, Villejuif
- Germany (5):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Italy (2):
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Turin, Piedmont
- GSK Investigational Site, Amsterdam, Netherlands
- Portugal (2):
  - GSK Investigational Site, Cascais
  - GSK Investigational Site, Lisbon
- Spain (2):
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Seville
- United Kingdom (4):
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Brighton, Sussex East
  - GSK Investigational Site, Birmingham, Warwickshire
  - GSK Investigational Site, London